CLINICAL TRIAL: NCT05019313
Title: Diaphragm Ultrasound Evaluation During Weaning From Mechanical Ventilation in the Positive COVID-19 Patient
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Luigi Vetrugno, Clinical Professor in Anesthesiology and Intensive Care, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: COVID-DIAUS 1.2
Record Dates: First submitted 2021-08-02; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: COVID-19 Pneumonia; Diaphragm Disease
Keywords: diaphragm thickening fraction; happy hypoxemia; diaphragmatic ultrasound evaluation; SARS-CoV-2 pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID 19 positive patients: COVID19 positive patients with hypoxemic acute respiratory failure hospitalized in intensive care unit.
  This study evaluates diaphragmatic contractility with ultrasound, blood gas analytical parameters during weaning from invasive mechanical ventilation
  Interventions: Device: Evaluation of diaphragmatic contractility by ultrasound

INTERVENTIONS:
Device: Evaluation of diaphragmatic contractility by ultrasound — Lung ultrasound is performed during mechanical ventilation weaning. The diaphragmatic thickening fraction is evaluated positioning a linear probe in midaxillary line. Inspiratory and expiratory measurements are bilateral and are M-mode images. Right diaphragmatic thickening fraction has been considered as true and reproducible measurement.

SUMMARY:
Hypoxemic acute respiratory failure is one of the main COVID-19 patients complication that lead to in intensive care hospitalization.

This complication determines a variable mortality from 25 to 30%. To correct hypoxemia (often severe) is often needed non-invasive or invasive mechanical ventilation.

Mechanical ventilation is not a therapeutic strategy, but it allows to extend the time-to-recovery necessary to solve COVID-19 respiratory failure cause.

Calibration of ventilatory support is essential to ensure adequate time-to-recovery without contributing to onset lung and / or diaphragmatic damage.

Basal diaphragmatic activity assessment, device for administering the oxygenation support choice and setting ventilatory support parameters are decisive.

Ultrasound is the best method for measuring diaphragmatic work. The aim of this study is to evaluate the diaphragmatic thickening fraction in COVID-19 patients admitted to Intensive Care Unit (ICU) for acute respiratory failure and to record its function on weaning.

DETAILED DESCRIPTION:
Hypoxemic acute respiratory failure in COVID-19 patients often leads to necessity of intubation and mechanical ventilation support. Complications may be severe as Ventilator-Induced Lung Injury (VILI) and respiratory infections. Weaning process from mechanical ventilation is based on respiratory work reduction and mechanical support to allow patient's respiratory ability to recovery. Respiratory muscle strength give an important contribute. Ultrasound diaphragmatic evaluation is essential to evaluate patients respiratory capacity as diaphragm atrophy usually suggest a difficult process and weaning failure.

COVID-19 pneumonia represent a particular type of ARDS (acute respiratory distress syndrome), in which different mechanism such as interstitial edema and diffuse alveolar damage, ventilation-perfusion mismatch, intrapulmonary shunt play a role/attend The aim of this study is to assess diaphragmatic function in weaning from mechanical ventilation in patients affected from COVID-19 respiratory failure and his implications.

ELIGIBILITY:
Inclusion Criteria:

* Hypoxemic respiratory failure in COVID-19 patients during intensive care unit hospitalization
* Age> 18 years
* Weaning by mechanical ventilation

Exclusion Criteria:

* tracheostomy,
* unstable clinical conditions;
* agitation (Richmond Agitation-Sedation Scale (RASS)≥ + 2) or non-cooperation (Kelly Matthay scale ≥5);
* more than two organ failure
* consent refusal

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe hypoxemic covid-related respiratory failure admitted to intensive care unit in Udine and five other centers. These subjects required mechanical ventilation during hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic function evaluation by measuring right diaphragmatic thickening fraction | During weaning by mechanical ventilation before attempt of extubation
  Right diaphragmatic thickening fraction is evaluated by positioning a linear ultrasound probe at the level of the midaxillary line (pointer oriented towards the axillary cavity). Patient is in the supine position. Inspiratory and expiratory measurements are made as M-mode images. Right diaphragmatic measurement is considered as a reference. .

SECONDARY OUTCOMES:
Weaning attempt success/failure frequency with consequent need of tracheostomy or endotracheal re-intubation. | After weaning and eventually extubation
  After extubation it is considered as weaning attempt success a 48 hours time free need of non invasive (not prophylatic) or invasive ventilation with re-intubation and/or tracheostomy

OTHER OUTCOMES:
Duration of mechanical ventilation. | from intubation to the end of mechanical ventilation support
  hours record/assessment of mechanical ventilation after intubation
ICU and Hospital length of stay and mortality. | from first day of hospitalization (admission to the hospital) to the last day (discharge from the hospital), an average of 90 days
  number of days in ICU and hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Intensive Care Clinic - Department of Medicine - ASUIUD, Udine, Italy

REFERENCES:
- [Background] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Background] Azoulay E, Thiery G, Chevret S, Moreau D, Darmon M, Bergeron A, Yang K, Meignin V, Ciroldi M, Le Gall JR, Tazi A, Schlemmer B. The prognosis of acute respiratory failure in critically ill cancer patients. Medicine (Baltimore). 2004 Nov;83(6):360-370. doi: 10.1097/01.md.0000145370.63676.fb. PMID 15525848
- [Background] Thiery G, Azoulay E, Darmon M, Ciroldi M, De Miranda S, Levy V, Fieux F, Moreau D, Le Gall JR, Schlemmer B. Outcome of cancer patients considered for intensive care unit admission: a hospital-wide prospective study. J Clin Oncol. 2005 Jul 1;23(19):4406-13. doi: 10.1200/JCO.2005.01.487. PMID 15994150
- [Background] Gattinoni L, Chiumello D, Caironi P, Busana M, Romitti F, Brazzi L, Camporota L. COVID-19 pneumonia: different respiratory treatments for different phenotypes? Intensive Care Med. 2020 Jun;46(6):1099-1102. doi: 10.1007/s00134-020-06033-2. Epub 2020 Apr 14. No abstract available. PMID 32291463
- [Background] Vetrugno L, Bove T, Orso D, Barbariol F, Bassi F, Boero E, Ferrari G, Kong R. Our Italian experience using lung ultrasound for identification, grading and serial follow-up of severity of lung involvement for management of patients with COVID-19. Echocardiography. 2020 Apr;37(4):625-627. doi: 10.1111/echo.14664. Epub 2020 Apr 15. PMID 32239532
- [Derived] Vetrugno L, Orso D, Corradi F, Zani G, Spadaro S, Meroi F, D'Andrea N, Bove T, Cammarota G, De Robertis E, Ferrari S, Guarnieri M, Ajuti M, Fusari M, Grieco DL, Deana C, Boero E, Franchi F, Scolletta S, Maggiore SM, Forfori F. Diaphragm ultrasound evaluation during weaning from mechanical ventilation in COVID-19 patients: a pragmatic, cross-section, multicenter study. Respir Res. 2022 Aug 21;23(1):210. doi: 10.1186/s12931-022-02138-y. PMID 35989352